CLINICAL TRIAL: NCT06850207
Title: Effect of Anticoagulant and Antiplatelet Drug Intervention on Postoperative Major Adverse Events in Patients with Peripheral Arterial Disease：Phase II
Brief Title: Effect of Anticoagulant and Antiplatelet Drug Intervention on Postoperative Major Adverse Events in Patients with PAD：Phase II
Status: Not yet recruiting | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, Chief Physician, Chengdu University of Traditional Chinese Medicine
Other Study IDs: ChengduUTCM11
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Disease(PAD)
Keywords: peripheral arterial disease; Anticoagulant and Antiplatelet Drug; Adverse Events
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is a multicenter, prospective, observational research project. It is anticipated to enroll a total of 6,000 patients between February 1, 2025, and January 31, 2028 (with completion of one-year postoperative follow-up by January 31, 2029). Patients will be grouped according to different combinations of anticoagulant and antiplatelet drugs used postoperatively for PAD. The types, dosages, and duration of postoperative anticoagulant and antiplatelet drug use will be recorded. Follow-up assessments will be conducted at 1 month, 6 months, and 12 months postoperatively to document the occurrence of Major Adverse Cardiovascular Events (MACE) and Major Adverse Limb Events (MALE) in the enrolled patients.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) refers to a group of chronic ischemic conditions caused by arterial intimal thickening, calcification, and secondary thrombus formation, leading to arterial stenosis or even occlusion. It is a localized manifestation of systemic atherosclerotic disease. The condition often affects the distal abdominal aorta and large to medium-sized arteries such as the iliac, femoral, and popliteal arteries, and may extend to distal main arteries like the popliteal artery in advanced stages. Clinical manifestations range from mild to severe, including cold limbs, fatigue after walking, intermittent claudication, rest pain, ulcers, and necrosis. PAD predominantly affects middle-aged and elderly individuals, and its incidence continues to rise due to population aging and dietary changes, reaching 15%-30% among those aged 70. It has become one of the most common diseases in vascular surgery.

Revascularization can rapidly restore blood flow and alleviate limb ischemia symptoms, but it does not fundamentally address the chronic, systemic, and progressive nature of atherosclerosis in PAD patients. The risk of cardiovascular and lower limb vascular events remains. Studies have shown that the risk of acute limb ischemia increases fourfold after lower limb arterial revascularization, while the risk of myocardial infarction rises by 30%. Therefore, while endovascular therapy quickly improves limb symptoms, efforts should be made to actively reduce the risk of cardiovascular and limb events.

In 2017, the European Society for Vascular Surgery (ESVS) emphasized the importance of antiplatelet therapy after revascularization in PAD patients, although the recommendation was based on Class C evidence. From 1982 to 1991, six retrospective studies demonstrated that aspirin effectively improves graft patency rates. The 2000 BOA study found that warfarin doubled the risk of major bleeding after PAD surgery, with no significant benefits except for reducing venous graft occlusion. The 2010 CASPAR study showed that dual antiplatelet therapy with clopidogrel and aspirin also doubled the risk of bleeding. In 2018, the VOYAGER study revealed that for high-risk limb ischemia patients, rivaroxaban combined with aspirin reduced the incidence of vascular events compared to aspirin monotherapy. In the same year, the COMPASS study demonstrated that for high-risk cardiovascular ischemic events, the combination of rivaroxaban and aspirin effectively reduced cardiovascular event rates without increasing bleeding risk.

Data from the Vascbase database indicate that in real-world practice, postoperative antithrombotic treatments are not limited to rivaroxaban and aspirin. Various drug combinations are used, but their safety and efficacy remain unverified. Therefore, in 2023, Professor Wu Ziheng from the Vascular Surgery Department of the First Affiliated Hospital of Zhejiang University School of Medicine initiated a clinical study titled "The Impact of Anticoagulant and Antiplatelet Drug Interventions on Postoperative Adverse Events in Patients with Peripheral Arterial Disease," abbreviated as "The Coach-PAD Study" (ClinicalTrials.gov Identifier: NCT05852197). This study aims to explore the effects of different anticoagulant and antiplatelet drug combinations on cardiovascular and lower limb events after PAD surgery, providing high-level evidence from real-world data for postoperative antithrombotic therapy in PAD patients. By December 2024, nearly 7,000 participants had been enrolled. Due to data capacity limitations in the Vascbase database, the study is being extended. Thus, our center is launching the second phase of the clinical study, "The Impact of Anticoagulant and Antiplatelet Drug Interventions on Postoperative Adverse Events in Patients with Peripheral Arterial Disease," to further investigate the effects of different anticoagulant and antiplatelet drug combinations on cardiovascular and lower limb events after PAD surgery.### Research Content

* 1. Study Population Patients undergoing endovascular treatment for lower extremity arteriosclerosis obliterans.
* 2. Participant Selection Criteria

  1. Patients diagnosed with lower extremity arteriosclerosis obliterans and undergoing endovascular treatment;
  2. Patients who voluntarily sign the informed consent form.
* 3. Sample Size Calculation This is a prospective real-world study with minimal enrollment criteria, employing non-probability sampling. The sample size estimation is based on the Vascbase database, which records approximately 2,500 patients annually. Therefore, the goal is to recruit 6,000 patients with lower extremity arterial disease over three years.
* 4. Specific Research Content Patients will be grouped according to different combinations of anticoagulant and antiplatelet drugs used postoperatively for PAD. The types, dosages, and duration of postoperative anticoagulant and antiplatelet drug use will be recorded. Follow-up assessments will be conducted at 1 month, 6 months, and 12 months postoperatively to document the occurrence of Major Adverse Cardiovascular Events (MACE) and Major Adverse Limb Events (MALE).

  ### Research Methods
* 1. Enrollment Criteria (Diagnostic Criteria, Inclusion Criteria, Exclusion Criteria) **1.1 Diagnostic Criteria:**

  1. Typical clinical manifestations of lower extremity arteriosclerosis obliterans, such as intermittent claudication, rest pain, toe ulcers, or gangrene;
  2. Physical examination revealing weakened or absent distal arterial pulses;
  3. Imaging studies (e.g., ultrasound, CT, MRI, or DSA) confirming stenosis or occlusion of lower extremity arteries.

**1.2 Inclusion Criteria:**

1. History of PAD or intermittent claudication, with an ankle/brachial index (ABI) < 0.9 or angiography-confirmed significant peripheral arterial stenosis (≥50%);
2. Undergoing endovascular treatment for aortoiliac, femoral, popliteal, or infrapopliteal arteries;
3. No restrictions on endovascular treatment methods, including all internationally recognized devices and techniques used in real-world practice;
4. Willingness to sign the informed consent form.

**1.3 Exclusion Criteria:**

1) History of stroke within the past month or hemorrhagic/lacunar stroke; 2) Known ejection fraction < 30% or severe heart failure with Class III/IV symptoms; 3) Non-cardiovascular diseases associated with poor prognosis (e.g., metastatic cancer) or interventions that increase the risk of adverse events; 4) History of allergies or contraindications to rivaroxaban, aspirin, or other study drugs; 5) Known liver diseases associated with coagulation disorders; 6) Pregnancy, lactation, or women of childbearing potential who are sexually active and not using effective contraception; 7) Contraindications to any study-related procedures.

* 2. Participant Grouping Patients will be grouped based on different combinations of anticoagulant and antiplatelet drugs used postoperatively.
* 3. Criteria for Early Withdrawal/Termination

  1. Voluntary withdrawal of informed consent by the patient;
  2. Other circumstances deemed necessary by the investigator for withdrawal.

     * Study Procedures
* 1. Participant Management

  1. **Recruitment Methods:** Suitable patients will be recruited during clinical practice.
  2. **Informed Consent Process:** Clinical researchers will educate patients and obtain informed consent.
  3. **Verification of Inclusion/Exclusion Criteria:** Clinical researchers will verify enrollment criteria.
  4. **Review of Medical History and Concomitant Medications:** Clinical researchers will review and record medical history and concomitant medications.
* 2. Safety Evaluation Procedures (Adverse Event Assessment, Monitoring, and Reporting) As an observational study, this research does not influence patient treatment and thus does not impose additional risks. Any adverse events occurring during treatment will be managed by the attending physician according to clinical guidelines. Researchers will promptly document adverse events and their outcomes.
* 3. Risk Control and Management Procedures

  * **Drug and Device Standards:** All devices and drugs used must be approved by the National Medical Products Administration and included in the hospital's fee schedule.
  * **Monitoring Plan:** Before enrollment, the study sponsor will assess the rationality of diagnoses and collect data through the system. Monitoring will include verifying the completeness of in-hospital data, addressing issues, and making corrections as needed.
  * **Study Closure Phase:** After completing in-hospital records, patients will undergo regular online and offline follow-ups to ensure clear and complete documentation.
* 4. Visit Requirements

The expected follow-up period is 12 months. Based on published literature and clinical experience, the study will proceed as follows:

1. **Screening Phase:**

   * Pre-enrollment visit (-10 to -1 day): Patients sign informed consent, complete medical history, including vital signs, symptoms, past medical history, general and preoperative tests (e.g., CBC, liver function, renal function, coagulation profile, lipid panel, ECG).
2. **Treatment Phase:**

   * Baseline visit (day of surgery, day 0): Record vital signs, symptoms, surgical details, and evaluate treatment efficacy and adverse events.
3. **Post-Treatment Visits (Safety Follow-Up, Follow-Up, Survival Follow-Up):**

   * Postoperative visit (1 to 21 days post-surgery): Quality of life assessment, record concomitant medications, and document adverse events.
   * Follow-up 1 (1 month ± 7 days): Quality of life assessment, record concomitant medications, and document adverse events.
   * Follow-up 2 (6 months ± 30 days): Quality of life assessment, record concomitant medications, and document adverse events.
   * Follow-up 3 (12 months ± 30 days): Quality of life assessment, record concomitant medications, and document adverse events.

     ### Study Start and End
   * **Recruitment:** February 2025 to January 2028, aiming to enroll 6,000 patients undergoing endovascular treatment for lower extremity arteriosclerosis obliterans.
   * **Follow-Up:** February 2025 to January 2029, completing 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* 1. History of PAD, or a history of intermittent claudication with an ankle/brachial blood pressure ratio < 0.9, or angiography-confirmed significant peripheral arterial stenosis (≥50%).

  2. Underwent endovascular treatment for aortoiliac, femoral, popliteal, or infrapopliteal arteries.

  3. No restrictions on endovascular treatment methods, including all internationally recognized devices and techniques used in real-world practice.

  4. Agreed and signed the informed consent form.

Exclusion Criteria:

* 1. **Patients with a history of stroke within the past month** or a history of hemorrhagic or lacunar stroke.

  2. Patients with a known ejection fraction < 30% or severe heart failure with Class III/IV symptoms.

  3. Patients with non-cardiovascular diseases associated with poor prognosis(e.g., metastatic cancer) or interventions that increase the risk of adverse events in the study.

  4. Patients with a history of allergies or known contraindications to drugs such as rivaroxaban or aspirin.

  5. Patients with any known liver disease associated with coagulation disorders. 6. Pregnant or breastfeeding women, or women of childbearing potential who are sexually active and not using effective contraception.

  7. Patients with known contraindications to any study-related procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing endovascular treatment for lower extremity arteriosclerosis obliterans
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Composite Adverse Event Rate (MACE/MALE): Myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation due to vascular disease. | From enrollment to the end of treatment at 12 months
  MACE (Major Adverse Cardiovascular Events):
  Includes acute myocardial infarction, severe arrhythmia, heart failure, ischemic stroke, and death. Follow-up and recording will be conducted at 1 month, 6 months, and 12 months postoperatively.
  MALE (Major Adverse Limb Events):
  Includes major amputation, bleeding events (such as cerebral hemorrhage and gastrointestinal bleeding), and reintervention of the ipsilateral lower limb artery. Assessments will be performed at 1 month, 6 months, and 12 months postoperatively.

SECONDARY OUTCOMES:
MACE（Major Adverse Cardiovascular Events） | From enrollment to the end of treatment at 12 months
  MACE (Major Adverse Cardiovascular Events):
  Includes acute myocardial infarction, severe arrhythmia, heart failure, ischemic stroke, and death. Follow-up and recording will be conducted at 1 month, 6 months, and 12 months postoperatively

OTHER OUTCOMES:
MALE（Major Adverse Limb Events） | From enrollment to the end of treatment at 12 months
  MALE (Major Adverse Limb Events):
  Includes major amputation, bleeding events (such as cerebral hemorrhage and gastrointestinal bleeding), and reintervention of the ipsilateral lower limb artery. Assessments will be performed at 1 month, 6 months, and 12 months postoperatively.
Composite Freedom from Vascular Adverse Events | From enrollment to the end of treatment at 12 months
  Composite Freedom from Vascular Adverse Events refers to the absence of any of the aforementioned events (MACE, MALE, or major bleeding) during the follow-up period.
All-Cause Mortality | From enrollment to the end of treatment at 12 months
  All-cause mortality refers to death from any cause.

IPD SHARING:
Plan to Share IPD: No